CLINICAL TRIAL: NCT06836336
Title: Effectiveness of Digital Versus Hybrid Interventions in Promoting Nutrition Knowledge Among Adolescent Girls: A Randomized Trial
Brief Title: Digital Versus Hybrid Interventions in Promoting Nutrition Knowledge Among Saudi Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Essra Noorwali, Associate Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HAPO-02-K-012-2023-10-1787
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Nutrition Knowledge; Generalized Anxiety Disorder (GAD); Food Habits; Body Mass Index
Keywords: Diet; Anxiety; Nutritional knowledge; Educational intervention; Saudi Arabia; Adolescents; Digital; Hybrid intervention
MeSH Terms: conditions — Generalized Anxiety Disorder; Feeding Behavior; Anxiety Disorders | interventions — Hybrid Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to one of two groups. First group received a hybrid intervention that combined face-to-face educational sessions with the integration of technological advancements. They attended weekly 40-minute interactive educational sessions over the course of a month. The educational materials encompass information regarding the components of a healthy balanced diet and an active lifestyle. This content was developed by a professional team, including registered dietitians and physicians. Second group received a fully digital intervention, they received the same educational materials through WhatsApp twice a week over the course of one month. The educational materials were presented through easily understandable posters, brief videos, and followed by short quizzes to reinforce the acquired knowledge. The digital intervention incorporated the same behavior change strategies that were utilized in the hybrid group. Participants were introduced to MyFittnessPal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid intervention (Experimental): Hybrid intervention that combined face-to-face educational sessions with the integration of technological advancements.
  Interventions: Behavioral: Hybrid therapy
- Fully digital intervention (Experimental): Received the same educational materials as the hybrid intervention group through WhatsApp twice a week over the course of one month.
  Interventions: Behavioral: Fully digital

INTERVENTIONS:
Behavioral: Hybrid therapy — Hybrid intervention that combined face-to-face educational sessions with the integration of technological advancements. They attended weekly 40-minute interactive educational sessions over the course of a month. The educational materials encompass information regarding the components of a healthy balanced diet and an active lifestyle.Throughout the intervention, participants were provided with a range of behavior change techniques to support participants in applying the educational content to improve their dietary and lifestyle habits. The employed behavior change techniques were SMART (specific, measurable, achievable, relevant, time-bound) goal setting, reviewing behavioral goals, problem-solving and environmental restructuring. The technological support for this intervention included the use of a smartphone diet tracker app called MyFitneesPal as well as communication with the interventionists via WhatsApp.
  Arms: Hybrid intervention
Behavioral: Fully digital — Fully digital intervention, where they received the same educational materials through WhatsApp twice a week over the course of one month. The educational materials were presented through easily understandable posters, brief videos, and followed by short quizzes to reinforce the acquired knowledge. Additionally, the digital intervention incorporated the same behavior change strategies that were utilized in the hybrid group. Participants were also introduced to MyFittnessPal application in order to help them track their dietary habits and monitor their progress since it is considered a tool for self-monitoring and promoting healthy dietary behaviors throughout the intervention period.
  Arms: Fully digital intervention

SUMMARY:
This study primarily aims to compare the efficacy of different approaches to nutrition education intervention delivery in improving nutrition knowledge (NK) among Saudi adolescent girls. A secondary aim is to compare the effectiveness of these interventions in enhancing dietary habits and reducing Generalized Anxiety Disorder (GAD) scores.A randomized sample of 104 Saudi adolescent girls aged 16-18 years from a single high school in Makkah city enrolled in a 4-week lifestyle educational intervention for health promotion. Participants were randomly assigned to either a hybrid or a fully digital nutritional education program. Outcome measures included knowledge (NK), dietary and lifestyle habits assessed by the Healthy Plate Variety Score (HPVS), and mental health evaluated using the Generalized Anxiety Disorder (GAD) scores.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Adolescents (15-19 years old)
* Reliable internet access
* Willing to participate

Exclusion Criteria:

* Has chronic disease/s
* <15 years and >19 years
* No internet access
* Not willing to participate

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Nutrition knowledge | From enrollment to the end of treatment at 4 weeks
  Nutritional Knowledge was assessed using a validated dietary questionnaire, distributed in Arabic (24). The questionnaire comprised 10 items, with a maximum score of 10 points. Each correct response was awarded 1 point, while incorrect answers or uncertain responses received a score of zero. The final score was derived by summing the total points. To classify NK levels, modified Bloom's cut-off points were employed: a score of 80-100% (8-10 points) indicated good NK, 50-79% (5-7.9 points) represented moderate knowledge, and scores below 50% (<5 points) denoted low knowledge. For analytical purposes, these categories were dichotomized into satisfactory NK (>80% correct) and unsatisfactory NK (<80% correct) (7,25).

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Scores (GAD) | From enrollment to the end of treatment at 4 weeks
  Anxiety levels were measured using the GAD-7. This is a 7-item validated questionnaire (28), which is widely used to screen for and quantify the severity of GAD. The Arabic version of this tool has been adopted by the Saudi Arabian Ministry of Health for initial anxiety screening. Each item is rated on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. Higher scores reflect greater anxiety levels. Anxiety was defined using a cutoff score of 10 or above, which differentiated between minimal to mild anxiety and moderate to severe anxiety (28).
Dietary habits | From enrollment to the end of treatment at 4 weeks
  Dietary habits were evaluated using a questionnaire adapted from research on food consumption frequencies in Qatar, which share similar characteristics with Saudi Arabia. The questionnaire assessed the frequency of consumption of various food groups, including vegetables, fruits, carbohydrates (e.g., bread, rice, pasta), proteins (e.g., chicken, beef, fish), and dairy products (e.g. yoghurt and cheese). Participants responded to questions such as, "How often do you consume fresh fruits/green leafy vegetables/fish? To evaluate dietary variety, the study employed the Healthy Plate Variety Score, calculated using a modified methodology based on Jones et al. (2015). This approach involved dichotomizing food intake from the five main groups into two categories (daily intake vs. non-daily). Foods consumed daily received a score of 1, while those not consumed daily received a score of 0 with a potential maximum score of 5.0.
Anthropometric measurements (Body mass index) | From enrollment to the end of treatment at 4 weeks
  Body measurements were obtained using standardized equipment following established operating procedures. Trained senior dietitians objectively assessed the height and weight of adolescents using a mechanical combined scale and a stadiometer (Detecto). Prior to measurement, a technician ensured that the equipment was properly calibrated. Height was recorded to the nearest 0.1 cm while participants were barefoot and dressed in minimal clothing. Weight was measured and documented to the nearest 0.1 kg. The Body Mass Index (BMI) was calculated by dividing the weight in kilograms by the square of the height in meters. Weight status was classified according to the criteria set by the World Health Organization (WHO): underweight was defined as a BMI of less than 18.5 kg/m², normal weight ranged from 18.5 to 24.9 kg/m², overweight was categorized as a BMI between 25.0 and 29.9 kg/m², and obesity was indicated by a BMI of 30.0 kg/m² or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Mai A Ghabashi, PhD, Principal Investigator — Umm Al-Qura University
Locations (1):
- Al-Fatat Private School, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashton LM, Sharkey T, Whatnall MC, Williams RL, Bezzina A, Aguiar EJ, Collins CE, Hutchesson MJ. Effectiveness of Interventions and Behaviour Change Techniques for Improving Dietary Intake in Young Adults: A Systematic Review and Meta-Analysis of RCTs. Nutrients. 2019 Apr 11;11(4):825. doi: 10.3390/nu11040825. PMID 30979065
- [Background] Charles Shapu R, Ismail S, Ahmad N, Lim PY, Abubakar Njodi I. Systematic Review: Effect of Health Education Intervention on Improving Knowledge, Attitudes and Practices of Adolescents on Malnutrition. Nutrients. 2020 Aug 13;12(8):2426. doi: 10.3390/nu12082426. PMID 32823548
- [Background] Bany-Yasin H, Elmor AA, Ebrahim BK, Ahmed AAM, Alarachi MR, Abedalqader L, Amer R, Alyousef AMS, Alhajeh YF, Alyoussef A, Eid HAMA, Elsayed MM, Desouky EDE, Salem HK, Salem MR. Exploration of the nutrition knowledge among general population: multi-national study in Arab countries. BMC Public Health. 2023 Jun 19;23(1):1178. doi: 10.1186/s12889-023-15791-9. PMID 37337137
- [Background] Saha S, Okafor H, Biediger-Friedman L, Behnke A. Association between diet and symptoms of anxiety and depression in college students: A systematic review. J Am Coll Health. 2023 May-Jun;71(4):1270-1280. doi: 10.1080/07448481.2021.1926267. Epub 2021 Jun 4. PMID 34087087
- [Background] Lwin EZ, Watthanakulpanich D, Phetrak A, Soonthornworasiri N, Prangthip P. Factors influencing secondary school students' nutrition, mindfulness, and academic performance in Nan Province, Thailand. PLoS One. 2025 Jan 14;20(1):e0308882. doi: 10.1371/journal.pone.0308882. eCollection 2025. PMID 39808604
- [Background] Das JK, Salam RA, Thornburg KL, Prentice AM, Campisi S, Lassi ZS, Koletzko B, Bhutta ZA. Nutrition in adolescents: physiology, metabolism, and nutritional needs. Ann N Y Acad Sci. 2017 Apr;1393(1):21-33. doi: 10.1111/nyas.13330. PMID 28436102
- [Background] Hargreaves D, Mates E, Menon P, Alderman H, Devakumar D, Fawzi W, Greenfield G, Hammoudeh W, He S, Lahiri A, Liu Z, Nguyen PH, Sethi V, Wang H, Neufeld LM, Patton GC. Strategies and interventions for healthy adolescent growth, nutrition, and development. Lancet. 2022 Jan 8;399(10320):198-210. doi: 10.1016/S0140-6736(21)01593-2. Epub 2021 Nov 29. PMID 34856192
- [Background] Hamulka J, Czarniecka-Skubina E, Gutkowska K, Drywien ME, Jeruszka-Bielak M. Nutrition-Related Knowledge, Diet Quality, Lifestyle, and Body Composition of 7-12-Years-Old Polish Students: Study Protocol of National Educational Project Junior-Edu-Zywienie (JEZ). Nutrients. 2023 Dec 19;16(1):4. doi: 10.3390/nu16010004. PMID 38201834

DOCUMENTS (1):
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT06836336/ICF_000.pdf